CLINICAL TRIAL: NCT04432870
Title: Patients' Preferences About Rescheduling Colonoscopies Delayed Due to COVID-19: Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of the Health Decision Sciences Center, Massachusetts General Hospital
Other Study IDs: 2020P001579-1
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Colon Cancer
Keywords: shared decision making; colon cancer screening; COVID-19; waitlist
MeSH Terms: conditions — Colonic Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MGH Patients: Patients aged 45-75 who had their screening or surveillance colonoscopy postponed or delayed due to the COVID pandemic at Massachusetts General Hospital

SUMMARY:
The study is a cross-sectional survey study targeting patients aged 45-75 who had their screening or surveillance colonoscopy postponed or delayed due to the COVID pandemic. Study staff will survey a random subsample of patients to assess anxiety, COVID risk tolerance, cancer worry, willingness to screen and barriers to screening colonoscopy, and preference for colonoscopy and alternative colon cancer screening options.

Eligible patients will be sent a survey packet in the mail that will include a cover letter, an information sheet describing the study, an incentive, and the survey. The cover letter will include information for participants to opt-out if they desire. Patients will be asked to complete the survey and return it back to study staff. Consent is implied with return of the survey.

For the study, staff plan to invite 300 patients and expect to receive 195 completed surveys. Analyses will examine whether COVID-19 has changed patients' interest in colon cancer screening and the strength of patients' preferences for colonoscopy and other approaches to colon cancer screening. It will then examine factors associated with positive and negative views on rescheduling colonoscopies such as anxiety, worry, and risk perceptions.

DETAILED DESCRIPTION:
The study is a cross-sectional survey study targeting patients aged 45-75 who had their screening or surveillance colonoscopy postponed or delayed due to the COVID pandemic. Staff will survey a random subsample of patients to assess anxiety, COVID risk tolerance, cancer worry, willingness to screen and barriers to screening colonoscopy, and preference for colonoscopy and alternative colon cancer screening options.

Study staff will work with the gastroenterology department to identify patients whose colonoscopy has been delayed due to COVID-19 and who meet the eligibility criteria. A random sample of about 300 eligible patients will be selected for the survey study.

Eligible patients will be sent a survey packet in the mail that will include a cover letter, an information sheet describing the study, an incentive, and the survey. The cover letter will include information for participants to opt-out if they desire. Patients will be asked to complete the survey and return it back to study staff. Patients will also be able to complete the survey online via a RedCap link. Consent is implied with return of the completed survey. Staff will make up to three reminder phone calls and will send a reminder packet to non responders.

The study staff will invite 300 patients and expect to receive about 195 completed surveys.

Analyses will first examine whether there are differences between responders and non responders. Then, the analysis will examine descriptive statistics exploring patients' interest in colon cancer screening, strength of preference for switching to stool based testing or postponing colonoscopy for a year. The analyses will explore patients' perspective towards colonoscopy in the coming months and factors associated with positive or negative perceptions of colonoscopy such as anxiety, cancer worry, COVID worry and risk perceptions. The relationships between these factors will be examined using chi-square analysis (for categorical data) and correlations (for continuous data). Models will be used to explore factors associated with different preferences for screening.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 45-75
* Had screening or surveillance colonoscopy delayed due to COVID-19
* Either first screening colonoscopy or a routine screening or surveillance colonoscopy for low to moderate risk patients (as indicated by 3-10 year recommended follow up frequency from prior test)

Exclusion Criteria:

* Diagnostic colonoscopy
* High risk for colorectal cancer as indicated by 1 year follow up schedule
* Prior history of colon cancer or irritable bowel syndrome
* Unable to read or write in English or Spanish

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 45-75 who had their colonoscopy delayed or postponed due to the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Interest in colon cancer screening | at start of study--between one week and 2 months after start of study
  Item with 5-point response assessing whether COVID-19 has increased, decreased or not changed interest in colon cancer screening

SECONDARY OUTCOMES:
Preference for stool testing | at start of study--between one week and 2 months after start of study
  Item with 5-point response (definitely want to definitely do not want) measuring interest in having a stool test for colon cancer
Preference for postponing colonoscopy for one year | at start of study--between one week and 2 months after start of study
  Item with 5-point response (definitely want to definitely do not want) measuring interest in postponing colonoscopy for one year
Worry about delay | at start of study--between one week and 2 months after start of study
  Item with 5 point response (extremely worried to not at all worried) assessing worry about the delay of the colonoscopy on their colon cancer risk
Risk perception on COVID-19 | at start of study--between one week and 2 months after start of study
  Item with 5-point response (very high to very low) assessing patients' perception about risk of getting COVID-19 from having a colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To promote research replicability, transparency and future use of the data, de-identified data sets of the patient survey data will be created and will be available, by request, to outside researchers.
  After the main manuscripts have been published, de-identified data sets will also be deposited in an open access service such as, ICPSR (https://www.icpsr.umich.edu/icpsrweb/). Before a dataset is made available for access, ICPSR completes a detailed review of all datasets to assess disclosure risk. If necessary, ICPSR modifies data to reduce disclosure risk or limits access to datasets for which modifying the data would substantially limit their utility or the risk of disclosure remains high. No information that contains identifiers or that could be used to link an individual to the data will be included in the de-identified data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Three months after the end of the funded grant period, the study materials and de-identified data will be available, by request, from the PI. Once data are placed on an open access service such as ICPSR they will be available indefinitely.
Access Criteria: The PI will share a de-identified data set with outside investigators at no cost, according to approved Partners and Massachusetts General Hospital policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.
  On ICPSR, individuals must register and agree to ICPSR's Responsible Use statement prior to accessing datasets.